CLINICAL TRIAL: NCT04111848
Title: Evaluation of the Effect of Adding Magnesium Sulfate Infusion to Ketamine Infusion on Improvement of the Analgesic Efficacy in Cancer Breast Surgeries.
Brief Title: Magnesium and Ketamine in Postoperative Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AP1904-50102
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Analgesia
Keywords: Magnisum sulfate; Ketamine; Analgesia; Breast Cancer Surgeries
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Magnesium

STUDY DESIGN:
Intervention Model Description: 90 female patients scheduled for cancer breast surgeries will be assigned to 2 groups, each of 45. Group (K) will receive a bolus of 0.5 mg/kg ketamine with induction of anaesthesia, followed by ketamine infusion 0.12 mg/kg/hour continued till 24 hours after surgery. Group (KM) will receive a bolus of 0.5 mg/kg ketamine added to 50mg/kg magnesium sulfate over 30 minutes after induction of anaesthesia, followed by ketamine infusion 0.12 mg/kg/hour added to 8mg/kg/hour of magnesium sulfate continued till 24 hours after surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study medications were prepared by a pharmacist who was not involved in the patient management or the data collection. Both the patients and the stuff involved in their management were unaware of the group assignment. Equal rates of the drug infusion and equal volumes of the administered drugs were applied to all patients to ensure double blinding of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ketamine group : group (k) (Experimental): -Ketamine group (group K): will receive a bolus of 0.5 mg/kg ketamine during induction of anaesthesia diluted in 100 ml normal saline, followed by ketamine infusion 0.12 mg/kg/hour continued till 24 hours after surgery. The infusion pump concentration will be 0.6mg/ml and the rate of infusion will be 0.2 ml/kg/hour
  Interventions: Drug: Ketamine
- ketamine and magnesium group: group (KM) (Experimental): - Ketamine and magnesium group (group KM): will receive a bolus of 0.5 mg/kg ketamine added to 50mg/kg magnesium sulfate diluted in 100 ml normal saline over 30 minutes after induction of anaesthesia, followed by ketamine infusion 0.12 mg/kg/hour added to 8mg/kg/hour of magnesium sulfate continued till 24 hours after surgery. Each ml of the administered infusion will contain 0.6mg ketamine and 40mg magnesium and the rate of infusion will be 0.2 ml/kg/hour.
  Interventions: Drug: ketamine and magnesium

INTERVENTIONS:
Drug: Ketamine — Patients will be assigned into 2 groups (each of 45):
  Ketamine group (group K): will receive a bolus of 0.5 mg/kg ketamine during induction of anaesthesia diluted in 100 ml normal saline, followed by ketamine infusion 0.12 mg/kg/hour continued till 24 hours after surgery. The infusion pump concentration will be 0.6mg/ml and the rate of infusion will be 0.2 ml/kg/hour.
  Arms: ketamine group : group (k)
Drug: ketamine and magnesium — Ketamine and magnesium group (group KM): will receive a bolus of 0.5 mg/kg ketamine added to 50mg/kg magnesium sulfate diluted in 100 ml normal saline over 30 minutes after induction of anaesthesia, followed by ketamine infusion 0.12 mg/kg/hour added to 8mg/kg/hour of magnesium sulfate continued till 24 hours after surgery. Each ml of the administered infusion will contain 0.6mg ketamine and 40mg magnesium and the rate of infusion will be 0.2 ml/kg/hour.
  Arms: ketamine and magnesium group: group (KM)

SUMMARY:
90 female patients scheduled for cancer breast surgeries will be assigned to 2 groups, each of 45. Group (K) will receive a bolus of 0.5 mg/kg ketamine with induction of anaesthesia, followed by ketamine infusion 0.12 mg/kg/hour continued till 24 hours after surgery. Group (KM) will receive a bolus of 0.5 mg/kg ketamine added to 50mg/kg magnesium sulfate over 30 minutes after induction of anaesthesia, followed by ketamine infusion 0.12 mg/kg/hour added to 8mg/kg/hour of magnesium sulfate continued till 24 hours after surgery. The same anaesthetic regimen will be applied to all patients. Total intraoperative fentanyl required to maintain mean blood pressure within 20% of its baseline will be recorded. After surgery, all patients will be connected to PCA device containing morphine solution, the amount of morphine consumed during the first 24 hours will be recorded. In the follow-up visits after 3 months, all patients will be assessed for neuropathic pain by DN4 questionnaire.

DETAILED DESCRIPTION:
90 female patients aged between 18 and 65 years, scheduled for cancer breast surgeries will be assigned to 2 groups, each of 45. Group (K) will receive a bolus of 0.5 mg/kg ketamine with induction of anaesthesia, followed by ketamine infusion 0.12 mg/kg/hour continued till 24 hours after surgery. Group (KM) will receive a bolus of 0.5 mg/kg ketamine added to 50mg/kg magnesium sulfate over 30 minutes after induction of anaesthesia, followed by ketamine infusion 0.12 mg/kg/hour added to 8mg/kg/hour of magnesium sulfate continued till 24 hours after surgery. The same anaesthetic regimen will be applied to all patients. Total intraoperative fentanyl required to maintain mean blood pressure within 20% of its baseline will be recorded. After surgery, all patients will be connected to PCA device containing morphine solution, the amount of morphine consumed during the first 24 hours will be recorded. In the follow-up visits after 3 months, all patients will be assessed for neuropathic pain by DN4 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with class II physical status (American Society of Anaesthesiologists) ,
* Age between 18-65 years,
* Scheduled for breast cancer surgery (e.g. modified radical mastectomy and conservative mastectomy)

Exclusion Criteria:

* Patient refusal,
* Cardiac dysfunction (ejection fraction <45%),
* Diabetic patients
* Patients with uncontrolled hypertension
* Patients have any degree of heart block
* Patients have renal impairment (creatinine > 2 mg/dl),
* Patients have hepatic dysfunction (transaminases > 2 times normal),
* Patients with preexisting neurological or psychiatric disease,
* Patients who are allergic to one of the study drugs,
* Patients with communication difficulties,
* Inability to use the patient controlled analgesia (PCA) device,
* Female patients who are pregnant
* Patients who use preoperative calcium channel blockers or narcotic drugs.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
the total amount of morphine required during the first postoperative 24 hours | the first postoperative 24 hours
  After transferring to post-anaesthesia care unit (PACU), the IV route of each patient will be connected to a PCA device containing morphine solution (1mg/ml). This PCA device will be set to deliver a demand dose of 1ml with a lockout interval of 15 minutes and without a continuous background infusion.
  The primary outcome in this study will be assessed in the form of the total amount of morphine required during the first postoperative 24 hours.

SECONDARY OUTCOMES:
the total amount of intraoperative fentanyl consumption | during anaesthesia (intraoperative)
  the total amount of intraoperative fentanyl required to maintain values of mean blood pressure within 20% of their baseline values
(Visual Analogue scale) VAS scores | the first postoperative 24 hours
  (VAS) scores during rest and with shoulder movement at 0, 4, 8, 12and 24 post-operative hours
Douleur Neuropathique 4 (DN4 | 3 months after surgery
  Chronic post-operative pain will be evaluated in all patients during their outpatient follow-up visit after 3 months. Patients with score of ≥ 4 in the Douleur Neuropathique 4 (DN4) questionnaire will indicate the incidence of neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hassan, MD, Principal Investigator — Ass Prof- Anesthesia Dept- National Cancer Institute - Cairo University
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassan ME, Mahran E. Effect of magnesium sulfate with ketamine infusions on intraoperative and postoperative analgesia in cancer breast surgeries: a randomized double-blind trial. Braz J Anesthesiol. 2023 Mar-Apr;73(2):165-170. doi: 10.1016/j.bjane.2021.07.015. Epub 2021 Jul 29. PMID 34332956